CLINICAL TRIAL: NCT06113328
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of MK-6194 in Adult Participants With Non-Segmental Vitiligo
Brief Title: A Clinical Study of MK-6194 for the Treatment of Vitiligo (MK-6194-007)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6194-007; 2023-503502-37-00 (Registry Identifier: EU CT); U1111-1287-4329 (Registry Identifier: UTN); MK-6194-007 (Other: MSD); jRCT2031230622 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Non-segmental Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Base Study: Dose 1 (Experimental): Participants receive subcutaneous (SC) MK-6194 dose regimen 1.
  Interventions: Biological: MK-6194
- Base Study: Dose 2 (Experimental): Participants receive SC MK-6194 dose regimen 2.
  Interventions: Biological: MK-6194; Drug: Placebo
- Base Study: Placebo (Placebo Comparator): Participants receive an SC placebo regimen.
  Interventions: Drug: Placebo
- Extension: Dose 1 (Experimental): Participants receive SC MK-6194 dose regimen 1. Participants from the arms "Base Study: Dose 1" or "Base Study: Placebo" may be enrolled in this arm after completing participation in their original arm.
  Interventions: Biological: MK-6194
- Extension: Dose 2 (Experimental): Participants receive SC MK-6194 regimen 2. Participants from the arms "Base Study: Dose 2" or "Base Study: Placebo" may be enrolled in this arm after completing participation in their original arm.
  Interventions: Biological: MK-6194; Drug: Placebo

INTERVENTIONS:
Biological: MK-6194 — MK-6194 administered subcutaneously (SC)
  Arms: Base Study: Dose 1; Base Study: Dose 2; Extension: Dose 1; Extension: Dose 2
Drug: Placebo — Placebo comparator to MK-6194 administered SC
  Arms: Base Study: Dose 2; Base Study: Placebo; Extension: Dose 2

SUMMARY:
Researchers are looking for a new way to treat people with non-segmental vitiligo (NSV). The goal of this study is to learn about the safety of MK-6194 and how well people tolerate it. Researchers also want to learn if people who take MK-6194 have more of a decrease in the amount of vitiligo on their face compared to people who take placebo.

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of non-segmental vitiligo
* Has non-segmental vitiligo with disease duration of at least 6 months
* Has depigmentation contributing to Facial Vitiligo Area Scoring Index (F-VASI) ≥ 0.3 at screening and baseline
* Has depigmented facial body surface area (BSA) ≥0.3% at screening and baseline
* Has Total Vitiligo Area Scoring Index (T-VASI) ≥4 at screening and baseline
* Has total body vitiligo area ≥4% at screening and baseline excluding hands and feet involvement

Exclusion Criteria:

* Has segmental vitiligo
* Has ≥50% leukotrichia on face or body
* Has any other dermatological diseases that would interfere with vitiligo assessments
* Has history of or current inflammatory condition other than vitiligo that, in the opinion of the investigator, could interfere with the evaluation of vitiligo
* Has a known systemic hypersensitivity to interleukin 2 (IL-2), or modified IL-2 including MK-6194, or its inactive ingredients
* Has an active or clinically significant infection requiring hospitalization or treatment with IV anti-infectives within 4 weeks prior to Randomization, or oral/intramuscular anti-infective therapy within 2 weeks prior to Randomization
* Has symptomatic heart failure (New York Heart Association class III or IV) or myocardial infarction or unstable angina pectoris within 6 months prior to Screening
* Has a severe chronic pulmonary disease requiring oxygen therapy
* Has a transplanted organ, which requires continued immunosuppression
* Has a history of any malignancy, except for successfully treated non-melanoma skin cancer or localized carcinoma in situ of the cervix
* Has evidence of active tuberculosis (TB), latent TB, or inadequately treated TB
* Has confirmed or suspected COVID-19 infection
* Has history of drug or alcohol abuse within 6 months prior to Screening
* Has had major surgery within 3 months prior to Screening OR has a major surgery planned during the study
* Has had an inadequate response (as evaluated by a dermatologist or local physician specialist equivalent) to previous treatment with a Janus kinase inhibitor (JAKi) after an appropriate treatment duration (eg, ≥12 weeks)
* Has received prohibited medications within protocol-specified timeframes prior to Randomization
* Has participated in another investigational clinical study within 4 weeks prior to Randomization
* Has donated or lost ≥1 unit of blood (approximately 500 mL) within 4 weeks prior to the Screening Visit
* Has received cosmetic or other procedures that could interfere with evaluation of vitiligo during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Facial Vitiligo Area Scoring Index (F-VASI) at Week 24 | Baseline and Week 24
  VASI is a validated scoring method that assesses the extent and severity of areas of vitiligo depigmentation. F-VASI will be calculated to indicate facial lesions, using the following scale: At 100% depigmentation, no pigment is present; at 90%, specks of pigment are present; at 75%, the depigmented area exceeds the pigmented area; at 50%, the depigmented and pigmented areas are equal; at 25%, the pigmented area exceeds the depigmented area; and at 10%, only specks of depigmentation are present.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 24 weeks
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 24 weeks
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Change from Baseline in Total Vitiligo Area Scoring Index (T-VASI) at Week 24 | Baseline and Week 24
  VASI is a validated scoring method that assesses the extent and severity of areas of vitiligo depigmentation. T-VASI will be calculated to indicate all lesions on the body, using the following scale: At 100% depigmentation, no pigment is present; at 90%, specks of pigment are present; at 75%, the depigmented area exceeds the pigmented area; at 50%, the depigmented and pigmented areas are equal; at 25%, the pigmented area exceeds the depigmented area; and at 10%, only specks of depigmentation are present.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (68):
- United States (13):
  - Cahaba Dermatology & Skin Health Center ( Site 0127), Birmingham, Alabama
  - Burke Pharmaceutical Research ( Site 0124), Hot Springs, Arkansas
  - The Vitiligo & Pigmentation Institute of Southern California ( Site 0115), Los Angeles, California
  - Indiana University Health University Hospital-Indiana University School of Medicine, Department of (, Indianapolis, Indiana
  - Dawes Fretzin Clinical Research Group, LLC ( Site 0106), Indianapolis, Indiana
  - Metro Boston Clinical Partners ( Site 0110), Brighton, Massachusetts
  - Hamzavi Dermatology - Canton ( Site 0101), Canton, Michigan
  - Remington Davis Clinical Research-Outpatient ( Site 0104), Columbus, Ohio
  - Medical University of South Carolina-Dermatology Research ( Site 0114), Charleston, South Carolina
  - International Clinical Research - Tennessee LLC ( Site 0120), Murfreesboro, Tennessee
  - Progressive Clinical Research ( Site 0108), San Antonio, Texas
  - Virginia Clinical Research, Inc. ( Site 0109), Norfolk, Virginia
  - Dermatology Specialists of Spokane ( Site 0126), Spokane, Washington
- Argentina (5):
  - Psoriahue ( Site 0205), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Stat Research S.A. ( Site 0204), Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Metabólicas (CINME)-Dermatology ( Site 0203), Buenos Aires, Buenos Aires F.D.
  - Instituto Medico Strusberg ( Site 0208), Córdoba, Córdoba Province
  - Hospital Aleman-Dermatologia ( Site 0209), Buenos Aires
- Australia (4):
  - Paratus Clinical Research Woden ( Site 1703), Phillip, Australian Capital Territory
  - Westmead Hospital-Dermatology ( Site 1701), Westmead, New South Wales
  - Skin Health Institute Inc.-Trials ( Site 1702), Carlton, Victoria
  - Sinclair Dermatology ( Site 1704), Melbourne, Victoria
- Belgium (2):
  - UZ Gent ( Site 0604), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0601), Leuven, Vlaams-Brabant
- Canada (4):
  - Enverus Medical Research ( Site 0006), Surrey, British Columbia
  - Diex Recherche Quebec Inc. ( Site 0008), Québec, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain ( Site 0002), Québec, Quebec
  - Diex Recherche sherbrooke Inc. ( Site 0007), Sherbrooke, Quebec
- Chile (5):
  - Dermisur ( Site 0305), Osorno, Los Lagos Region
  - Clinical Research Chile SpA ( Site 0304), Valdivia, Los Ríos Region
  - Clinica Dermacross ( Site 0301), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-CICUC ( Site 0308), Santiago, Region M. de Santiago
  - Centro Internacional de Estudios Clinicos (CIEC) ( Site 0302), Santiago, Region M. de Santiago
- Colombia (5):
  - CliniSalud ( Site 0401), Envigado, Antioquia
  - IPS SURA San Diego ( Site 0408), Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe ( Site 0405), Barranquilla, Atlántico
  - Healthy Medical Center S.A.S ( Site 0403), Zipaquirá, Cundinamarca
  - Fundación Valle del Lili ( Site 0412), Cali, Valle del Cauca Department
- France (4):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet ( Site 0803), Nice, Alpes-Maritimes
  - CHU de Bordeaux Hop St ANDRE ( Site 0804), Bordeaux, Aquitaine
  - Hôpital Edouard Herriot ( Site 0802), Lyon, Auvergne-Rhône-Alpes
  - HENRI MONDOR HOSPITAL ( Site 0801), Créteil, Val-de-Marne
- Germany (3):
  - Universitaetsklinikum Erlangen-Hautklinik Studienambulanz ( Site 0905), Erlangen, Bavaria
  - Universitätsklinikum Münster-Hautklinik ( Site 0904), Münster, North Rhine-Westphalia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0901), Berlin
- Israel (2):
  - Rambam Health Care Campus-Dermatology ( Site 1002), Haifa
  - Sheba Medical Center-Dermatology ( Site 1001), Ramat Gan
- Japan (3):
  - Nagoya City University Hospital-Dermatology ( Site 2002), Nagoya, Aichi-ken
  - Osaka University Hospital ( Site 2004), Suita, Osaka
  - Tokyo Medical University Hospital ( Site 2001), Shinjuku-ku, Tokyo
- Mexico (3):
  - Cryptex Investigación Clínica S.A. de C.V. ( Site 0515), Cuauhtémoc, Ciudad de México, Mexico City
  - Unidad biomedica avanzada monterrey-Clinical Trials ( Site 0504), Monterrey, Nuevo León
  - Centro de Atención e Investigación Clínica ( Site 0507), Aguascalientes
- Amsterdam UMC, locatie AMC-Dermatology ( Site 1101), Amsterdam, North Holland, Netherlands
- South Korea (3):
  - Inha University Hospital ( Site 1992), Incheon
  - Seoul National University Hospital-Dermatology ( Site 1991), Seoul
  - Severance Hospital, Yonsei University Health System-Department of Dermatology ( Site 1993), Seoul
- Spain (3):
  - Hospital Universitario Puerta del Mar ( Site 1302), Cadiz, Andalusia
  - Hospital Universitari de Bellvitge-Dermatology ( Site 1307), L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra ( Site 1305), Madrid, Madrid, Comunidad de
- Switzerland (2):
  - Cantonal Hospital St.Gallen ( Site 1402), Sankt Gallen, Canton of St. Gallen
  - UniversitätsSpital Zürich ( Site 1401), Zurich, Canton of Zurich
- Turkey (Türkiye) (3):
  - Hacettepe Universite Hastaneleri-Dermatology ( Site 1501), Altindağ, Ankara
  - Ankara Bilkent Şehir Hastanesi-Dermatology ( Site 1502), Ankara
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri-Dermatology and Venereology ( Site 1506), Kayseri
- United Kingdom (3):
  - Royal London Hospital-Dermatology Research Unit ( Site 1605), London, England
  - Queen Elizabeth Hospital Birmingham ( Site 1603), Birmingham, Warwickshire
  - New Cross Hospital ( Site 1601), Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26173&tenant=MT_MSD_9011